CLINICAL TRIAL: NCT03951272
Title: A Prospective, Multi-center, Randomized, Parallel-controlled Clinical Trial Evaluating the Efficacy and Safety of Lyoplant Onlay in Repairing Cerebral Dura Mater
Brief Title: The Efficacy and Safety of Lyoplant® Onlay in Repairing Cerebral Dura Mater
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: B. Braun Medical International Trading Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-G-H-1715
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Replacement and Extension of Connective Tissue Structure in Neurosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyoplant® Onlay (Experimental): All the model including 2.5cm×2.5cm, 5.0cm×5.0cm,2.5cm×7.5cm,7.5cm×7.5cm,10.0cm×12.5cm will be used in this study
  Interventions: Device: Lyoplant® Onlay/DURAFORM™ Dural Graft Implant
- DURAFORM™ Dural Graft Implant (Active Comparator): All the model including 2.54cm×2.54cm,5.08cm×5.08cm, 2.54cm×7.62cm, 7.62cm×7.62cm,10.16cm×12.70cm will be used in this study
  Interventions: Device: Lyoplant® Onlay/DURAFORM™ Dural Graft Implant

INTERVENTIONS:
Device: Lyoplant® Onlay/DURAFORM™ Dural Graft Implant — Lyoplant® Onlay will be used as a dura substitute for the repair of the duramater.The DURAFORM™ Dural Graft Implant will be used in the procedures where the repair or substitution of the patient's dura mater is needed.

SUMMARY:
Objective of this clinical trial is to compare the safety and efficacy of Mianfengxing Kexishou Yingmo Bupian(Lyoplant® Onlay) and Yingmo Bupianfor dural repair.270 subjects will be enrolled for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical patients who will receive dura mater replacement in neurosurgery;
2. 18 to 75 years old, either sexes;
3. Patients are ready and able to accept all visits during the trial.
4. Patients are willing and able to sign Informed Consent Form (ICF) to join this clinical trial.

Related to lesions:

1. Target lesion is cerebral and cerebellum dura mater defect closure, intracranial hypertension remission;
2. Surgical wound classification is Class I/sterile operation and risk index category (RIC) ≤ 2.

Exclusion Criteria:

1. Patients with local cerebral infection;
2. Patients who suffer from systemic infection (e.g. urinary tract infection (UTI), acquired pneumonia) or any infection sign at surgical site before the surgery, with body temperature > 38.5℃, positive result in blood culture, and/or positive result in chest X-ray examination;
3. Patients who are allergic to the equipment components (Such as, by asking the patient's history of allergies, doctors understand whether the patient is allergic to proteins of bovine origin or implant or not);
4. There is metal implant in patient's brain and the implant will interfere the assessment on devices or surgery recovery;
5. Patients in gestation period or lactation period or planned to be pregnant during the trial;
6. Patients with more than 1 separated dura mater defects;
7. Patients with previous neurosurgery history at the same anatomic site;
8. Patients with cranial open trauma;
9. Patients requiring the use of dura adhesive or sealant;
10. Patients whose expected survival time is less than 12 months;
11. Patients received chemotherapy and/or radiotherapy within 3 months before the surgery;
12. Patients who had diagnosed as malignant tumor of other parts except brain tumor, uncontrolled diabetes, septicemia, systemic collagen diseases clinically;
13. Patients who had been accompanied with liver and renal dysfunction, with ALT and AST>1.5 times the upper limit of the standard, total bilirubin level > 2.5 mg/dl, creatinine level > 2.0 mg/dl;
14. Patients with significant clinical coagulation disorders, Activated partial thromboplastin time (APTT) was 3 times more than ULN (upper limit of normal), international normalized ratio (INR) is ≥ 1.7, or under the treatment of Warfarin or Coumadin;
15. Patients with immune system damage or autoimmune diseases (white blood cell (WBC) count is < 4000/uL or >20,000/uL);
16. Patients whose serological test results show that people with hepatitis B, hepatitis C, syphilis, AIDS and other infectious diseases during screening period;
17. Patients in whom subdural drainage for more than 2 days must be performed in the surgery;
18. Patients who are participating other clinical trials of investigational devices/drugs;
19. Patients who are not suitable for this study as determined by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Surgical successful rate without leakage of cerebrospinal fluid (CSF) 90 days | 90days
  Surgical successful rate without leakage of cerebrospinal fluid (CSF) 90 days after the surgery (Confirmed by radiological image evaluation and physical examination on surgical site). Each patient firstly undergoes an initial CT and if necessary, MRI will be used to further examine the volume of CSF leakage.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No